CLINICAL TRIAL: NCT03692650
Title: Influence of Cognition and Physiological Function by Partial Sleep Deprivation of Taiwan University Students During Final Exam
Brief Title: Influence of Cognition and Physiological Function by Partial Sleep Deprivation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805059RINC
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-09

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Partial sleep deprivation (PSD), is a common problem among current university students in Taiwan. Students often get inadequate sleep time due to burden schoolwork during exam period. In recent years, Issue of sleep quality has gradually been emphasized. According to previous research, lacking in sleep easily results in sleepiness, fatigue, and poor problem-solving performance. Sleep deprivation may also affects cognitive performance, like reducing working memory performance. Furthermore, sleep deprivation will probably alter autonomic nervous function, such as sympathetic/parasympathetic activity change. Previous researches also suggested that sleep deprivation may associated with the risk of being obesity or suffering from diabetes. However, most researches focused on the effects of total sleep deprivation, especially those who usually have night shift work, such as medical staff. Few studies investigated the cognitive function and physiological function of university students after a period of time of partial sleep deprivation. As a results, the aim of the study is to investigate how partial sleep deprivation affects the cognitive performance and physiological function before and after the final exam period in healthy young university students between 20 and 30 years old in Taiwan, in order to promote the importance of healthy sleep and improve sleep quality among university students.

DETAILED DESCRIPTION:
40 healthy young university students who meet the inclusion criteria will be enrolled to the study. The investigators will detailed explain the research process to participants, and make sure all participants provide written informed consent. The study will be conducted in clinical cardiopulmonary function lab in school and graduate institute of physical therapy, college of medicine, National Taiwan University. Baseline evaluation will be conducted after all the midterm exam complete, and make sure there is no sleep deprivation events two weeks before and after baseline evaluation. Outcome measurement will be on the day after all final exams complete.

Participants will need to wear ActiGraph GT3X monitor (ActiGraph LLC, Pensacola, FL, USA), which is a non-invasive sleep monitoring device in order to record precise sleep hours and sleep condition, five days before baseline and outcome evaluation. On the days of both baseline and outcome evaluation, the investigators will provide computer device for participants to perform cognitive performance test, which will take around 15 minutes to complete. Next, participants can take a rest for 10 minutes on the bed in supine position before heart rate variability measurement starts. The investigators will place electrode on participant's right forearm, then the non-invasive device will record heart rate variability data for about 5 to 10 minutes. At last, the investigators will evaluate participant's dominant hand grasp strength (kg) by Jamar hand dynamometer (Jackson, MI, USA) devices in standing position.

ELIGIBILITY:
Inclusion Criteria:

* healthy young university students

Exclusion Criteria:

* People who cannot cooperate with the research
* Any medication that may affects the autonomic nervous system(such as beta blockers)
* Pregnancy
* People who have serious musculoskeletal/neurological/cardiopulmonary disorder or other systemic diseases that cannot complete the whole research tasks
* People who have already been diagnosed with any kinds of sleep disorders
* Without sleeping for more than 24 hours

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will recruit 40 healthy young university students between 20 to 30 years old as research participants
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
heart rate variability | Change from baseline heart rate variability at 4 weeks
  The investigator will use heart rate variation analyzer (SS1C,. Enjoy Research Inc., Taipei, Taiwan) to measure heart rate variability. Participant will lie on the bed in supine position, resting for 10 minutes before measurement. Baseline evaluation will be conducted on two weeks after all midterm exams completed and at least two months before the final exams starts. Outcome measurement will be on the first day after all final exams subjects complete.

SECONDARY OUTCOMES:
Grasp strength(kilogram) | Change from baseline grasp strength at 4 weeks
  The investigator will adopt Jamar hand dynamometer (Jackson, MI, USA) devices to evaluate dominant hand grasp strength(kg) of the participants. Each participant will perform 3 attempts maximal isometric muscle contractions in standing position and forearm neutral position, and the best performance will be recorded as an outcome. Baseline evaluation will be conducted on two weeks after all midterm exams completed and at least two months before the final exams starts. Outcome measurement will be on the first day after all final exams subjects complete.
Single N-back test(correct rate, %) | Change from baseline correct rate at 4 weeks
  Single n-back test will be used to evaluate working memory function and attention. The investigators will provide computer devices for all participants. Participants will perform 3 same tasks, each task spend 1 minutes. The average percentage of correct rate will be recorded as the outcome. Baseline evaluation will be conducted on two weeks after all midterm exams completed and at least two months before the final exams starts. Outcome measurement will be on the first day after all final exams subjects complete.
Stroop effects(seconds) | Change from baseline performance(seconds) at 4 weeks
  Stroop effects is widely used to evaluate attention, executive function, inhibition process, and automatic responses. The investigators will provide standard stroop charts(Traditional Chinese version) for all participants, which include 4 small parts in this charts. The investigators will record the time(seconds) of each parts that participant needs to complete as the outcome. Baseline evaluation will be conducted on two weeks after all midterm exams completed and at least two months before the final exams starts. Outcome measurement will be on the first day after all final exams subjects complete.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Yueh Chien, PhD, Study Chair — National Taiwan University, College of Medicine, Department of Physical Therapy
Locations (1):
- National Taiwan University, College of Medicine, Department of Physical Therapy, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patrick Y, Lee A, Raha O, Pillai K, Gupta S, Sethi S, Mukeshimana F, Gerard L, Moghal MU, Saleh SN, Smith SF, Morrell MJ, Moss J. Effects of sleep deprivation on cognitive and physical performance in university students. Sleep Biol Rhythms. 2017;15(3):217-225. doi: 10.1007/s41105-017-0099-5. Epub 2017 Apr 13. PMID 28680341
- [Background] Hirshkowitz M, Whiton K, Albert SM, Alessi C, Bruni O, DonCarlos L, Hazen N, Herman J, Katz ES, Kheirandish-Gozal L, Neubauer DN, O'Donnell AE, Ohayon M, Peever J, Rawding R, Sachdeva RC, Setters B, Vitiello MV, Ware JC, Adams Hillard PJ. National Sleep Foundation's sleep time duration recommendations: methodology and results summary. Sleep Health. 2015 Mar;1(1):40-43. doi: 10.1016/j.sleh.2014.12.010. Epub 2015 Jan 8. PMID 29073412
- [Background] Perez-Olmos I, Ibanez-Pinilla M. Night shifts, sleep deprivation, and attention performance in medical students. Int J Med Educ. 2014 Mar 29;5:56-62. doi: 10.5116/ijme.531a.f2c9. PMID 25341213
- [Background] Saadat H, Bissonnette B, Tumin D, Raman V, Rice J, Barry N, Tobias J. Effects of partial sleep deprivation on reaction time in anesthesiologists. Paediatr Anaesth. 2017 Apr;27(4):358-362. doi: 10.1111/pan.13035. Epub 2016 Nov 30. PMID 27900800
- [Background] Hershner SD, Chervin RD. Causes and consequences of sleepiness among college students. Nat Sci Sleep. 2014 Jun 23;6:73-84. doi: 10.2147/NSS.S62907. eCollection 2014. PMID 25018659
- [Background] Purim KS, Guimaraes AT, Titski AC, Leite N. Sleep deprivation and drowsiness of medical residents and medical students. Rev Col Bras Cir. 2016 Dec;43(6):438-444. doi: 10.1590/0100-69912016006005. English, Portuguese. PMID 28273216
- [Background] Tobaldini E, Costantino G, Solbiati M, Cogliati C, Kara T, Nobili L, Montano N. Sleep, sleep deprivation, autonomic nervous system and cardiovascular diseases. Neurosci Biobehav Rev. 2017 Mar;74(Pt B):321-329. doi: 10.1016/j.neubiorev.2016.07.004. Epub 2016 Jul 7. PMID 27397854
- [Background] Knutson KL, Spiegel K, Penev P, Van Cauter E. The metabolic consequences of sleep deprivation. Sleep Med Rev. 2007 Jun;11(3):163-78. doi: 10.1016/j.smrv.2007.01.002. Epub 2007 Apr 17. PMID 17442599
- [Background] Pasula EY, Brown GG, McKenna BS, Mellor A, Turner T, Anderson C, Drummond SPA. Effects of sleep deprivation on component processes of working memory in younger and older adults. Sleep. 2018 Mar 1;41(3). doi: 10.1093/sleep/zsx213. PMID 29361107
- [Background] Wang ML, Lin PL, Huang CH, Huang HH. Decreased Parasympathetic Activity of Heart Rate Variability During Anticipation of Night Duty in Anesthesiology Residents. Anesth Analg. 2018 Mar;126(3):1013-1018. doi: 10.1213/ANE.0000000000002439. PMID 29200073
- [Background] Nano MM, Fonseca P, Vullings R, Aarts RM. Measures of cardiovascular autonomic activity in insomnia disorder: A systematic review. PLoS One. 2017 Oct 23;12(10):e0186716. doi: 10.1371/journal.pone.0186716. eCollection 2017. PMID 29059210
- [Background] Zhong X, Hilton HJ, Gates GJ, Jelic S, Stern Y, Bartels MN, Demeersman RE, Basner RC. Increased sympathetic and decreased parasympathetic cardiovascular modulation in normal humans with acute sleep deprivation. J Appl Physiol (1985). 2005 Jun;98(6):2024-32. doi: 10.1152/japplphysiol.00620.2004. Epub 2005 Feb 17. PMID 15718408
- [Background] Lo JC, Ong JL, Leong RL, Gooley JJ, Chee MW. Cognitive Performance, Sleepiness, and Mood in Partially Sleep Deprived Adolescents: The Need for Sleep Study. Sleep. 2016 Mar 1;39(3):687-98. doi: 10.5665/sleep.5552. PMID 26612392
- [Background] Kuriyama K, Mishima K, Suzuki H, Aritake S, Uchiyama M. Sleep accelerates the improvement in working memory performance. J Neurosci. 2008 Oct 1;28(40):10145-50. doi: 10.1523/JNEUROSCI.2039-08.2008. PMID 18829972
- See also: Title: Lifestyle and Environmental Factors Associated with Sleep Quality of Preservice — http://www.airitilibrary.com/Publication/alDetailedMesh?docid=15618137-200806-x-52-1-11-a
- See also: Title: The Effects of Three Physical Trainings on Heart Rate Variability of the College Students after Sleep Deprivation — http://www.airitilibrary.com/Publication/alDetailedMesh?DocID=15610497-200812-8-3%264-77-84-a
- See also: Title: Sleep Deprivation and Fatigue in Clinicians — http://www.airitilibrary.com/Publication/alDetailedMesh?DocID=18102549-200603-3-3-194-200-a